CLINICAL TRIAL: NCT02047240
Title: Renal Function Determination With Creatinine and Cystatin C Dependent Formulas Compared to Gold Standard DTPA-TC-99 (Diethylene-triamine-pentaacetate- Technetium-99) in Mexican Cirrhotic Patients
Brief Title: Renal Function Determination in Patients With Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, Principal investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: FILT01
Record Dates: First submitted 2014-01-23; First posted 2014-01-28 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis; glomerular filtration; cystatin C
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
We have several ways to appropriately determine renal function in healthy patients and in several diseases, in cirrhotic population we dont have a precise tool that has sufficient precision that reflects glomerular function, although it has been reported that cystatin C, because of its nature could improve diagnostic accuracy to determinate the renal function in this population.

The investigators hypothesize that glomerular filtration obtained from cystatin-C-derived formulas are more accurate when compared to creatinine-derived formulas with DTPA-Tc99 (diethylene-triamine-pentaacetate- technetium-99) as gold standard.

DETAILED DESCRIPTION:
The aim of the study is to determine if the formulas for glomerular filtration are close to the estimation of actual renal function in mexican cirrhotic patients of different etiologies.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* Stability in creatinine levels in the previous three months (variation <0.3 mg/dL)
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Hepatocellular carcinoma
* Cerebrovascular events
* Decompensated heart failure
* Drugs that modify serum creatinine levels
* Renal replacement therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients will be selected from the Liver Clinic from the Gastroenterology Department at a tertiary care center in Mexico
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Levels of glomerular filtration through several formulas in cirrhotic patients | Baseline
  Determination of glomerular filtration through several formulas dependent of creatinine and cystatin C and the gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre, MD MSci, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", Mexico City, Mexico City, Mexico